CLINICAL TRIAL: NCT05213065
Title: Efficacy of Transnasal Sphenopalatine Ganglion Block Using TX360® Device for Children and Adolescents With Chronic Daily Headaches: A Single Center, Prospective, Randomized, Double Blind, Placebo-controlled Study Assessing the Efficacy of the Transnasal Sphenopalatine Ganglion Block in the Treatment of Chronic Daily Headache in Children and Adolescents
Brief Title: Assessment of the Efficacy of the Transnasal Sphenopalatine Ganglion Block in the Treatment of Chronic Daily Headache in Children and Adolescents.
Acronym: SPG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Pablo Ingelmo (Other)
Collaborators: Louise and Alan Edwards Foundation (Unknown)
Responsible Party: Sponsor-Investigator, Pablo Ingelmo, Head of Complex Pain Center ,Assistant Professor Pediatric-Anesthesiologist, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021-7715
Record Dates: First submitted 2021-05-20; First posted 2022-01-28 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Chronic Daily Headache; Post-Traumatic Headache
MeSH Terms: conditions — Headache Disorders; Post-Traumatic Headache | interventions — Sphenopalatine Ganglion Block; Bupivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Arm (Experimental): The participants randomized into this arm will receive the SPG block with 0.5% bupivacaine.
  Interventions: Other: Sphenopalatine ganglion block with 0.5% bupivacaine
- Placebo Arm (Placebo Comparator): The participants randomized into this arm will receive the SPG block with saline.
  Interventions: Other: Sphenopalatine ganglion block with saline

INTERVENTIONS:
Other: Sphenopalatine ganglion block with 0.5% bupivacaine — Repetitive SPG blockade using 0.5% bupivacaine delivered with the Tx360® device.
  Arms: Treatment Arm
Other: Sphenopalatine ganglion block with saline — Repetitive SPG blockade using saline delivered with the Tx360® device.
  Arms: Placebo Arm

SUMMARY:
Primary Objective The primary objective of the study is to assess whether transnasal sphenopalatine ganglion block using the device TX360 reduces intensity and severity of the Post-Traumatic Headache in adolescents.

Secondary Objectives

The study will also evaluate:

* Quality of life (QoL)
* Intensity of the headache
* Physical function
* Sleep quality
* Role function (measured by PEDMIDAS)
* Adverse events

DETAILED DESCRIPTION:
The sphenopalatine ganglion (SPG) is a large network of neurons that is easily accessible through the middle turbinate. The SPG is composed of branches from V1 and V2 of the trigeminal nerve and interconnects with sympathetic and parasympathetic autonomic fibers.6 The SPG has been successfully targeted transnasally to treat headache disorders and associated autonomic symptoms in adults.7 SPG blockade has been used in adults for treating several headache and facial pain conditions such as migraine, cluster headache, and trigeminal neuralgia.8 To our knowledge, there has not been any similar study done in children and adolescents.

The Tx360® device (Tian Medical Inc., Lombard, IL, USA) allows for noninvasive blockade of the SPG using a small catheter below the middle turbinate of the nose that is administered just beyond the pterygopalatine fossa. Regarding the efficacity of Tx360®, recent studies show that repetitive SPG blockade using 0.5% bupivacaine delivered with the Tx360® device was well-tolerated and effective at decreasing baseline headache intensity in adults.6

ELIGIBILITY:
Inclusion Criteria:

Subjects will be included if they meet all the following criteria:

1. Aged between 10 and 17.5 years old at the start of treatment
2. Daily Headache, within these categories:

   1. Persistent PTH attributed to Mild traumatic Brain injury to the head

Diagnostic criteria for persistent headache attributed to mild traumatic injury to the head:

Persistent headache attributed to traumatic injury to the head:

A. Any headache fulfilling criteria C and D B. Traumatic injury to the head1 has occurred

C. Headache is reported to have developed within 7 days after one of the following:

* Injury to the head
* Regaining of consciousness following injury to the head
* Discontinuation of medication(s) impairing ability to sense or report headache following injury to the head D. Headache persists for >3 months after its onset E. Not better accounted for by another ICHD-3 diagnosis Persistent headache attributed to mild traumatic injury to the head A. Headache fulfilling criteria for 5.2 Persistent headache attributed to traumatic injury to the head

B. Head injury fulfilling both of the following:

1. Associated with none of the following:

   * Loss of consciousness for >30 minutes
   * Glasgow Coma Scale (GCS) score <13
   * Post-traumatic amnesia lasting >24 hours1
   * Altered level of awareness for >24 hours
   * Imaging evidence of a traumatic head injury such as skull fracture, intracranial hemorrhage and/or brain contusion
2. Associated with one or more of the following symptoms and/or signs:

   * Transient confusion, disorientation or impaired consciousness
   * Loss of memory for events immediately before or after the head injury
   * Two or more of the following symptoms suggestive of mild traumatic brain injury:
   * Nausea
   * Vomiting
   * Visual disturbances
   * Dizziness and/or vertigo
   * Gait and/or postural imbalance
   * Impaired memory and/or concentration

Exclusion Criteria:

1. Previous history of brain imaging showing evidence of intracerebral hemorrhage, subdural or epidural hematomas, or subarachnoid hemorrhage as a consequence of traumatic head injury
2. Previous history of local anesthetic allergic reaction to bupivacaine
3. Nasal septal deformity or malformed facial or nasal passages such as cleft lip and palate, choanal atresia, atrophic rhinitis, rhinitis medicamentosa, septal perforation, deviation of the nasal septum, nasal/midface trauma or if he has recently had nasal/sinus surgery
4. Nasal or facial fracture impeding the use of TX360 device
5. Serious infection with congestion more than 10 days, and rectal temperature higher than 38°C for more than 1 day9.
6. Current diagnose of bleeding disorder or recurrent untreated (> 3/week) nosebleeds for the past 3 months
7. Severe respiratory distress, as noted by tachypnea or subcostal/intercostal retractions in when breathing
8. Angiofibroma, sinus tumors, or granuloma
9. Diagnosed or strongly suspected paroxysmal hemicrania or hemicrania continua
10. Pregnancy before the completion of the last dose
11. The possibility of a medication overuse headache is NOT an exclusion criterion, as long as the headache also corresponds to the inclusion criteria.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2022-02-05 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Number of Days of Headache per Month | up to 3 months after last intervention
  Number of Days of Headache per Month

SECONDARY OUTCOMES:
Pain Assessment during the headache | we will ask after every intervention and up to 3 months after last intervention
  using a Questionnaire that includes the following : Numerical Rating Scale (NRS), patients are asked to circle the number between 0 and 10, that fits best to their pain intensity . Zero usually represents 'no pain at all' whereas the upper limit represents 'the worst pain ever possible.
Patient Global Impression of Change scale ( PGIC) | asked in last visit and 1 month after last intervention again at 3 months after last intervention
  Patient Global Impression of Change scale ( PGIC) is a rating scale offered through a questionnaire that is most commonly used in clinically important changes after treatments and it has been used extensively in studies of musculoskeletal conditions. The patient is asked to describe changes in limitation, symptoms, emotions and overall quality of life related to the treatment received. Below is the scale that will be used:
  1. 'no change or condition got worse' = 0%;
  2. 'almost the same, hardly any change at all'=17%;
  3. 'a little better, but no noticeable change'=34%;
  4. 'somewhat better, but the change has not made any real difference'=50%;
  5. 'moderately better, and a slight but noticeable change' = 67%;
  6. 'better and definite improvement that has made a real and worthwhile difference
Measure Yourself Medical Outcome Profile ( MYMOP2) | Asked in : initial visit , visit 12 , 1 month post last intervention and 3 months after last intervention
  Measure Yourself Medical Outcome Profile (MYMOP2 ) is a 'patient-centred' outcome scale where patients are asked to nominate one or two symptoms (physical or mental) of a specific problem they need assistance with and consider the severity of these symptoms over the last week.
  Aims to measure the outcomes that the patient considers the most important. The patient chooses one or two symptoms for which they are seeking help and that they consider most important. They also choose an activity of daily living that is limited or prevented by these symptoms. These choices are written down in the patient's own words and the patient scores them for severity over the past week on a seven-point scale. Lastly, wellbeing is scored on a similar scale. On follow-up questionnaires, the wording of the previously chosen symptoms is unchanged. Follow-up questionnaires will be admin
Functional Disability Inventory(FDI) | Asked in : initial visit , visit 12 , 1 month post last intervention and 3 months after last intervention
  Functional Disability Inventory (FDI) was developed to measure physical functioning in school-aged children and adolescents. This measure relates to the ability to perform a range of everyday physical activities and has been well-established with different populations.
  The total FDI score is a sum of all of the items. Clinical reference points were developed to identify 3 categories of disability in pediatric chronic pain:
  * no/minimal disability (0 -12)
  * moderate disability (13-29)
  * severe disability (>30)
Pediatric Migraine Disability Assessment (PedMIDAS) | Asked in : initial visit , visit 12 , 1 month post last intervention and 3 months after last intervention
  Pediatric Migraine Disability Assessment (PedMIDAS) was developed to assess migraine disability in pediatric and adolescent patients
  It has been tested and validated for ages 4 to 18. The score is a simple composite of the total of six questions. If a range is provided, use the high end of the range or ask the family to provide a single number - both methods show equal validity. If the answer is blank or is a phrase (i.e., "few" or "couple"), they need to be asked to provide a number. The PedMIDAS grading scale is as follows:
  * Little or none disability (0-10)
  * Mild disability (11-30)
  * Moderate disability (31-50)
  * Severe disability (>50)
Pittsburgh Sleep Quality Index (PSQI) | Asked in : initial visit , visit 12 , 1 month post last intervention and 3 months after last intervention
  Pittsburgh Sleep Quality Index (PSQI) We evaluate sleep quality using PSQI. The scale counts 19 items assessing sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction. Point values of each item in of the seven subscales are summed and then combined as indicated to generate a subscale score. These totals are summed to create the global PSQI score. Scores range from 0-5 indicates good quality of sleep.
Number of Analgesic Medications used | up to 3 months after last intervention
  Patients will be encouraged to continue with their previous treatments and will not be asked to stop taking any medications in order to participate in this study. However, they will be allowed to reduce the doses or, eventually, to stop the use of analgesic medication under medical supervision.
  The number and class of analgesics taken will be collected at baseline, at the end of the treatment, and 1 and 3 months after the end of the treatment.
  The less the Analgesics medications used the Better .

OTHER OUTCOMES:
Number and Type of Adverse events | up to 3 months after last intervention
  By asking about side effects as :
  Dizziness, drowsiness, lacrimation, mouth numbness, throat, nasal irritation, bleeding, others.
  we will collect the number of side effects encountered as well as their severity .

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Ingelmo, MD, Principal Investigator — Research Institute at the Montreal Childrens Hospital
Locations (1):
- McGill University Health Centre (MUHC) - Montreal Children's Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kouri M, Somaini M, Cardenas VHG, Niburski K, Vigouroux M, Ingelmo P. Transnasal Sphenopalatine Ganglion Block for the Preventive Treatment of Chronic Daily Headache in Adolescents. Children (Basel). 2021 Jul 18;8(7):606. doi: 10.3390/children8070606. PMID 34356585